CLINICAL TRIAL: NCT06062979
Title: Clinical Effectiveness-Implementation Hybrid Type 2 Study on Home-Delivered Cabenuva for People Living With HIV Who Are Not Retained in Care
Acronym: CREATE
Status: Enrolling by invitation | Type: Observational
Sponsor: Whitman-Walker Institute (Other Government)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ViiV-219548
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: HIV
MeSH Terms: interventions — Rilpivirine; cabotegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Enhanced (MORE) implementation (i.e., MORE group): Study participants in this condition will be those engaged in clinical care as part of the MORE program, receiving supportive, wrap-around, and home-based HIV care services; all participants will be offered injectable Cabenuva and studied with regard to uptake and outcomes. Participants in this group will receive quantitative health survey assessments as per standard of care at Whitman-Walker Health. Participants will be offered quantitative and qualitative assessments regarding their experiences related to Cabenuva.
  Interventions: Drug: rilpivirine/cabotegravir
- Standard-of-care implementation (i.e., comparison group): Study participants in this comparison condition will be those engaged in clinical care receiving Cabenuva per standard of care at Whitman-Walker Health. Participants in this group will contribute ongoing electronic health record data under the auspices of an IRB-granted waiver of informed consent and waiver of HIPAA authorization.
  Interventions: Drug: rilpivirine/cabotegravir

INTERVENTIONS:
Drug: rilpivirine/cabotegravir — WWH is currently providing Cabenuva treatment as a treatment option for eligible patients. The purpose of the proposed study is to use an observational, prospective cohort design to further investigate the delivery of Cabenuva among two subpopulations of WWH patients.

SUMMARY:
The purpose of this study is to assess adherence to home-delivered long-acting injectable rilpivirine/cabotegravir (Cabenuva) among people living with HIV enrolled in the Mobile Outreach Retention and Engagement (MORE) program at Whitman-Walker Health due to significant barriers to being retained in care; the MORE program provides supportive services including dedicated care navigation, transportation assistance, and mobile/home-delivered care. The investigators will examine the equivalence of treatment outcomes among patients receiving injectable treatment within the MORE program as compared to those of patients receiving Cabenuva in standard care at Whitman-Walker Health.

DETAILED DESCRIPTION:
Advances in HIV treatment could promote better health and racial equity to address the gaps seen across the HIV care continuum nationally and locally. In Washington DC, HIV viral load suppression among People Living With HIV (PLWH) lies at 66%. Whitman-Walker Clinic, Inc., d/b/a Whitman-Walker Health (WWH), is a Federally Qualified Health Center ("FQHC") affiliated with Whitman-Walker Institute, Inc. ("Institute"). Institute is uniquely capable of addressing gaps with Cabenuva through WWH's existing MORE program, which includes supportive navigation and wrap-around services paired with home-based HIV care. However, there are many implementation knowledge gaps to identify with implementing Cabenuva injection protocols for PLWH who face significant barriers to retention in care and who may significantly benefit from integrating Cabenuva within the context of the MORE program.

The investigators propose a home-delivered Cabenuva HIV care program in Washington, D.C. to address the local HIV care continuum gaps. The investigative team has over five years of experience and lessons learned from our Mobile Outreach, Retention and Engagement (MORE) home-based HIV care program and plan to integrate Cabenuva therapy. MORE utilizes NP/PA providers and an HIV care navigator to deliver care to over 130 HIV-infected clients, who have a history of having fallen out of care, in their homes. The investigators envision that the inclusion of injectable treatment can expand the current program by geographic reach and the number of PWLH served by coupling Cabenuva with our ability to deliver patient-centered care outside of the traditional clinic. This proposal is critical to gathering early insights in Cabenuva implementation in Washington, D.C. and other EHE territories in FQHC clinic and affiliated non-clinic settings. Moreover, the data collected will demonstrate the extent to which a population experiencing significant barriers to retention in care-for whom Cabenuva would otherwise likely be counterindicated-can be supported via the MORE program to achieve comparable adherence and outcomes to typical patients receiving standard of care Cabenuva.

WWH is currently providing Cabenuva treatment as a treatment option for eligible patients. The purpose of the proposed study is to further investigate the delivery of Cabenuva among two subpopulations of WWH patients.

Cabenuva within standard clinical care at WWH: The majority of WWH patients receiving HIV treatment are offered and receive Cabenuva within the standard clinical setting. Among these patients, the proposed study will gather EMR-based data to characterize retention and HIV outcomes and to compare these and other relevant implementation factors with the MORE group. Medical providers identify eligible patients for Cabenvua based on a WWH protocol devised by medical leadership and a Cabenuva workgroup. Eligibility is viral load < 100,000 copies, no medication contraindications, no co-existing Hepatitis B infection, and no RAMs for rilpivirine or cabotegravir. Medical providers explain the risk and benefits and if the patient desires Cabeuva, the prescription is sent to the WWH onsite pharmacy at WWH sites MRC or 1525. The patient's case is sent via the EHR to the Cabenuva injection clinic admin lead at WWH. Patient appointment reminders and medication attainment are coordinated through SMS and phone call communication with patients.

Cabenuva within MORE-based clinical care at WWH: To address the unique structural and psychosocial factors that create significant barriers to engagement and retention in care for a subset of patients with a history of non-retention, the MORE program was developed. MORE's primary features include home-based care delivery, dedicated care navigation, transportation support, and wrap-around supportive services. WWH is currently expanding the MORE program to provide injectable Cabenuva to these patients for whom, without the intensive support of the MORE program, treatment with Cabenuva would likely be counterindicated. More follows a stepped-care approach to support that includes a customized combination of its services to each patient based on need and preferences.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals, aged 18 years or older, who are eligible to receive Cabenuva as standard of care at Whitman-Walker Health
* For those participants who will be prospectively enrolled via informed consent and offered survey and qualitative interviews, participants will be those receiving HIV-related treatment via the MORE program

Exclusion Criteria:

* HIV-uninfected individuals

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will be conducted among people living with HIV who are 18 years or older receiving HIV treatment at Whitman-Walker Health
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
4-month adherence rate | 4 months
  % of patients initiated who received each injection in the +/- 7 day window period for 4 months

SECONDARY OUTCOMES:
10-month adherence rate | 10 months
  % of patients who received each injection in the +/- 7 day window period for 10 months
Virologic suppression (200 copies/mL) | 1 through 12 months following first injection
  % of patients with virologic suppression (measured twice within 4 weeks and both values <200 copies/mL)
Virologic suppression (50 copies/mL) | 1 through 12 months following first injection
  % of patients with virologic suppression (measured twice within 4 weeks and both values <50 copies/mL)
Resistance associated viral mutations | 1 through 12 months following first injection
  % of patients with detection of resistance associated mutations

OTHER OUTCOMES:
Implementation Feasibility (qualitative) | 6 months
  Participants will be asked, "How easy was it to receive Cabenuva injections at home?"
Implementation Acceptability (qualitative) | 6 months
  Participants will be asked, "How do you like receiving an injection at home?"
Adoption Rate | 12 months
  # of providers who referred their patients to receive home-delivered Cabenuva among total number of providers

CONTACTS AND LOCATIONS:
Overall Officials: Megan Dieterich, PA, Principal Investigator — Whitman-Walker Institute
Locations (2):
- United States (2):
  - Whitman-Walker 1525 Clinic, Washington D.C., District of Columbia
  - Whitman-Walker Max Robinson Center, Washington D.C., District of Columbia